CLINICAL TRIAL: NCT02446808
Title: Clinical Assessment of Intraoperative Nerve Monitoring During Robot-assisted Laparoscopic Prostatectomy
Brief Title: Intraoperative Nerve Monitoring During Robot-assisted Laparoscopic Prostatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ProPep Surgical, LLC (Industry)
Collaborators: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ProPep B-016-001
Record Dates: First submitted 2015-05-11; First posted 2015-05-18 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Urinary Incontinence; Erectile Dysfunction
MeSH Terms: conditions — Urinary Incontinence; Erectile Dysfunction | interventions — Intraoperative Neurophysiological Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intraoperative nerve monitoring (Experimental): Patients for which intraoperative nerve monitoring (electromyography) is used to identify the location of somatic pelvic nerves critical to urinary continence control and erectile function in real time during robotic-assisted laparoscopic prostatectomy surgery
  Interventions: Device: Intraoperative nerve monitoring

INTERVENTIONS:
Device: Intraoperative nerve monitoring — Intraoperative nerve monitoring (electromyography) is used to identify the location of somatic pelvic nerves critical to urinary continence control and erectile function in real time during robotic-assisted laparoscopic prostatectomy surgery

SUMMARY:
The purpose of this study is to determine whether the use of intraoperative nerve monitoring during robotic-assisted laparoscopic prostatectomy surgery improves post-surgery urinary continence and erectile function.

DETAILED DESCRIPTION:
Study Design:

This is a single surgeon, single institution prospective post-market study of patients undergoing a robotic-assisted laparoscopic prostatectomy (RALP) with intraoperative nerve monitoring of pelvic nerves using the ProPep Nerve Monitoring System. The treatment group will consist of 80 subjects (with 69 anticipated to be evaluable) undergoing RALP with intraoperative nerve monitoring (IONM). This will be compared to a consecutive group of contemporary control cohort patients who have underwent RALP without nerve monitoring by the same single surgeon.

Baseline Evaluations and Data Collection:

Pre-operative baseline evaluations and data collection will be used to determine eligibility for enrollment and to document subject clinical status prior to surgical procedure. This information is recorded on the Screening case report forms (CRF).

The following data will be collected at screening/baseline:

* Medical History including Gleason score at biopsy, and clinical stage (cT, TNM 2002);
* Physical examination;
* Demographic information;
* Current symptoms;
* Expanded Prostate Cancer Index Composite for Clinical Practice (EPIC-CP) Questionnaire;
* SHIM Questionnaire;
* Use of any drugs for erectile dysfunction ;
* Confirmation of inclusion and exclusion criteria.

Surgical Procedure The surgical procedure should be completed according to site-specific standards. The following is a general overview of the surgical procedure for this study. The daVinci Surgical System must be used. Additional instrumentation necessary to perform the procedure is determined by the surgeon.

The Pep Electrode Introducer facilitates the introduction of the needle electrodes into the pelvis. The electrodes are initially placed in the levator muscle near the apex of the prostate in the area of the nerve bundles prior to the pedicle dissection to identify the perineal branches of the pudendal nerve. Prior to posterior dissection of the apex of the prostate, the needle electrodes are removed from the levator muscle and moved to the external urethral sphincter to identify the deep (muscular) branch of the perineal nerves. Action potentials are measured by the Pep Monitor.

Signals are induced in the nerve(s) of interest by stimulating the tissue surrounding the nerve(s) along the presumed nerve pathway with a low level electrical current. The low level current is delivered through the conventional bipolar instrument used during robotic surgery and when delivered close to a nerve it triggers and action potential in the nerve that is displayed on the Pep Monitor. The Pep Control Switch is used to switch the bipolar instrument between cautery mode and stimulation mode. The closer the bipolar instrument is to the nerve being located, the larger the amplitude of the action potential displayed by the Pep Monitor.

Nerves will be identified with the device prior to pedicle and apical dissection to establish nerve location. Nerve monitoring may be used through the course of dissections to confirm nerve location. Post-dissection readings will be collected after specimen removal to confirm the integrity of the preserved nerve tissue at the end of the case.

During the procedure and through hospital discharge the following data points will be collected:

* Type of nerve sparing - none, partial, and bilateral;
* Prostate size;
* Estimated blood loss and transfusion(s);
* Method of dissection (transperitoneal anterior, posterior, extraperitoneal, or lymph node dissection);
* Gleason score at radical prostatectomy;
* Pathological stage (nT);
* Positive surgical margin rate (PSM);
* Total robotic and surgical time;
* Total time for device deployment;
* Hospital admission / discharge dates; and
* Adverse events.

Postoperative care will be according to the site-specific standard of care.

Follow-up Evaluation and Data Collections:

Subjects will be followed post-operatively at catheter removal (typically 1 week), 1 month (±2 weeks), 3 months (±3 weeks), 6 months (±1 month), and 12 months (±1 month) following the procedure. Data will be collected on the appropriate follow-up Case Report Forms (CRFs). The CRFs for each of the follow-up data collection points will be supplied to the subjects upon their discharge from the hospital following their procedure. Research assistant will call subjects the week prior to the due date to remind subjects to fill in and mail back (via pre-addressed, stamped envelopes supplied with CRFs) appropriate CRF. Site specific standard of care will be followed post-operatively.

The following data and testing will be completed at each follow-up visit:

* Current symptoms;
* Modified EPIC-CP Questionnaire (question 3 and 4);
* SHIM Questionnaire;
* Use of any drugs for erectile dysfunction; and
* Adverse events (AE).

Contemporary Control Cohort:

As the procedures for the prospective cohort are standard of care at the investigators institution, the investigator will have all of the same measures for the contemporary control cohort that he has for the for the prospective cohort. Each prospective subject will be matched to two selected subjects in the contemporary control cohort by biopsy Gleason score (6 vs. 7 vs. 8-10), nerve-sparing status (yes/no), type of nerve sparing (unilateral or bilateral) and age (within 5 years). The contemporary control cohort will draw from consecutive patients who have undergone RALP in the previous two years (2012-2014) that did not have IONM. The investigator will not record AEs for this contemporary control cohort as the investigator is only interested in collecting AEs data potentially related to the use of the IONM.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects 40-70 years of age diagnosed with adenocarcinoma of the prostate;
* Subjects scheduled for robotic assisted radical prostatectomy for removal of localized prostate cancer;
* Subjects, who, in the opinion of the clinical Investigator, are able to understand this clinical investigation, cooperate with the investigational procedures and are willing to return for all the required post-treatment follow-up visits

Exclusion Criteria:

* Subjects with pre-operative urinary incontinence defined as use of pads or adult diapers;
* Subjects with previous pelvic or abdominal radiation therapy;
* Subjects with current or previous malignancy other than prostate or non-melanoma skin cancer;
* Subjects who have previously had a transurethral resection of the prostate (TURP) or holmium laser enucleation of the prostate (HoLEP), high intensity focused ultrasound (HIFU) or cryotherapy;
* Subjects with a prostate volume of >80mL
* Subjects with a body mass index (BMI) of ≥ 34;
* Subjects with current or suspected urinary tract or bladder infection(s);
* Subjects with reported unstable cardiovascular disease (e.g., unstable angina, myocardial infarction within past 6 months, cardiac failure or life-threatening arrhythmia, congestive heart failure) or symptomatic postural hypotension within 6 months before screening;
* Subjects with a history of diabetes;
* Subjects with drug, alcohol, or substance abuse reported within the last three years (subject reported);
* Subjects with a life expectancy less than study duration;
* Subjects with systemic autoimmune disorder;
* Subjects with any significant psychological disturbance that, in the opinion of the Investigator, could impair the consent process or ability to complete self-assessment questionnaires.
* Subjects with known sensitivity to any device or products required for the RALP surgery; and
* Subjects with any other condition that would contraindicate participation, as determined by the Investigator.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Return of urinary continence following robotic-assisted laparoscopic prostatectomy | 6 month
  The proportion of subjects who have urinary continence following robotic-assisted laparoscopic prostatectomy (RALP) at 6 months postoperatively.

SECONDARY OUTCOMES:
Return of erectile function following robotic-assisted laparoscopic prostatectomy | catheter removal which typically occurs at 1 week, 1 month, 3 month, 6 month, 12 month
  The proportion of subjects who return to pre-operative baseline (RTB) category (i.e. normal, mild, moderate, or severe erectile dysfunction) of erectile function following RALP with IONM of pelvic nerves. The change in SHIM score over time from baseline to 12 months.
Time to urinary continence | catheter removal which typically occurs at 1 week, 1 month, 3 month, 6 month, 12 month
  Assess time to continence defined as using 0 pads per day following RALP with IONM of pelvic nerves for 12 month post-operatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States